CLINICAL TRIAL: NCT05046340
Title: Applicability of Fluid Responsiveness Indices in Patients With Acute Circulatory Failure (AFRIC Study)
Brief Title: Applicability of Fluid Responsiveness Indices in Circulatory Failure (AFRIC Study) Study Project
Acronym: AFRIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Rui Shi, MD, PhD, Principal Investigator, Bicetre Hospital
Other Study IDs: 2017-A03580-53
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Shock; Acute Circulatory Failure
Keywords: pulse pressure variation; passive leg raising; end-expiratory occulsion test
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Passive leg raising — We perform the PLR test by adjusting the bed and not by manually raising the patient's legs. Bronchial secretions must be carefully aspirated before PLR. If awake, the patient should be informed of what the test involves. And measure the cardiac output by using certain devices at the bedside. The end-expiratory occlusion consists in interrupting the ventilator at end-expiration for 15-30 s and assessing the resulting changes in cardiac output.
  Other Names: end-expiratory occulsion test

SUMMARY:
Fluid administration is one of the main strategies for patients with acute circulatory failure. However, about half of the patients could not benefit from the fluid administration after the ICU admission. Thus predict the effect of fluid responsiveness is essential. There are sevral indices or tests can be used, such as pulse pressure variation (PPV), end-expiratory occulsion test (EEOT), passive leg raising (PLR), etc. Question of the prevalence of cases in which the different predictive indices of fluid responsiveness in intensive care unit (ICU) are not applicable.

DETAILED DESCRIPTION:
Fluid administration is one of the first-line therapies for most patients with acute circulatory failure. And it was supposed to increase cardiac preload and thus output significantly. However, it only has this effect if cardiac output is dependent on cardiac preload, that is if both ventricles work on the ascending part of the Frank-Starling curve. Our group had already shown that, in half of the critically ill patients admitted in ICU, fluid administration is likely to exert only deleterious effects without any hemodynamic benefit. To predict whether it will exert beneficial effects or not before administering the fluid therapy, a "dynamic approach" has been developed. It consists of observing the effects of changes of preload induced by various tests on cardiac output. 1) Pulse pressure variation: mechanical ventilation induces cyclical changes in cyclical changes in cardiac preload and right ventricular afterload due to cardiopulmonary interactions. If both ventricles are in a preload-dependent state, these variations will induce a cyclical variation in stroke volume. The latter being physiologically related to the pulsed arterial pressure (systolic - diastolic), the respiratory variation of the pulsed arterial pressure (PPV) indicates the existence of a preload-dependence of the two ventricles. 2) The End-expiratory occlusion test (EEOT): this is another method that takes advantage of heart-lung interactions to predict fluid responsiveness in ventilated patients. During mechanical ventilation, each insufflation increases intrathoracic pressure, which hinders systemic venous return. Thus, interrupting the respiratory cycle at the end of expiration inhibits this cyclic hindrance to venous return, increases cardiac preload and cardiac output if both ventricles are preload dependent. The duration of the EEOT must be at least 15 seconds. 3): Passive leg raising (PLR): when a patient is in a recumbent position, the elevation of the lower extremities and the horizontalization of the trunk passively transfers a significant volume of blood from the lower part of the body to the heart chambers and mimics volume expansion.

Numerous studies have reported that the increased cardiac output induced by PLR predicts fluid responsiveness. There is always the question of the prevalence of cases in which the different predictive indices of fluid responsiveness are not applicable and data on this issue are scarce, incomplete, and unsatisfactory.

Few studies have systematically investigated the number of patients in whom PPV cannot be used in the ICU settings. Some studies have reported a very low prevalence of cases where PPV was usable but they included the entire ICU population on a given day, including many patients who did not have an acute circulatory failure, which had no sense since PPV is only used in patients in whom the question of fluid therapy arises. Other studies have reported a higher prevalence of cases where PPV is usable, but they have only looked at the first 24 hours of hospitalization or have focused on patients with an unstable hemodynamic event. Finally, no study has ever studied the prevalence of cases where the respiratory variation of the PLR, or the EEOT are not applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. The presence of acute circulatory insufficiency defined by the following pragmatic criteria:

   * Prior administration of at least 1000 mL of crystalloid or colloid solute during a volemic expansion in the previous 12 hours
   * Norepinephrine administration/lactate ≥ 1.5 mmol/L

Exclusion Criteria:

* No strict exclusion criterion only if the refusal of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute circulatory failure need to evaluate fluid responsiveness.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of cases and reasons in which the conditions that the PPV cannot be correctly interpreted. | One minute at the bedside
  By using one arterial line, the scope at the bedside could have a PPV value that automatly calculated on the screen.
The prevalence of cases and reasons in which the conditions that the EEOT cannot be correctly interpreted. | 15 seconds for EEOT
The prevalence of cases and reasons in which the conditions that the PLR cannot be correctly interpreted. | One minute fot the passive leg raising

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benes J, Kirov M, Kuzkov V, Lainscak M, Molnar Z, Voga G, Monnet X. Fluid Therapy: Double-Edged Sword during Critical Care? Biomed Res Int. 2015;2015:729075. doi: 10.1155/2015/729075. Epub 2015 Dec 22. PMID 26798642
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Michard F, Boussat S, Chemla D, Anguel N, Mercat A, Lecarpentier Y, Richard C, Pinsky MR, Teboul JL. Relation between respiratory changes in arterial pulse pressure and fluid responsiveness in septic patients with acute circulatory failure. Am J Respir Crit Care Med. 2000 Jul;162(1):134-8. doi: 10.1164/ajrccm.162.1.9903035. PMID 10903232
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Heenen S, De Backer D, Vincent JL. How can the response to volume expansion in patients with spontaneous respiratory movements be predicted? Crit Care. 2006;10(4):R102. doi: 10.1186/cc4970. PMID 16846530
- [Background] Soubrier S, Saulnier F, Hubert H, Delour P, Lenci H, Onimus T, Nseir S, Durocher A. Can dynamic indicators help the prediction of fluid responsiveness in spontaneously breathing critically ill patients? Intensive Care Med. 2007 Jul;33(7):1117-1124. doi: 10.1007/s00134-007-0644-9. Epub 2007 May 17. PMID 17508201
- [Background] Muller L, Louart G, Bousquet PJ, Candela D, Zoric L, de La Coussaye JE, Jaber S, Lefrant JY. The influence of the airway driving pressure on pulsed pressure variation as a predictor of fluid responsiveness. Intensive Care Med. 2010 Mar;36(3):496-503. doi: 10.1007/s00134-009-1686-y. Epub 2009 Oct 22. PMID 19847400
- [Background] Malbrain ML, Reuter DA. Assessing fluid responsiveness with the passive leg raising maneuver in patients with increased intra-abdominal pressure: be aware that not all blood returns! Crit Care Med. 2010 Sep;38(9):1912-5. doi: 10.1097/CCM.0b013e3181f1b6a2. No abstract available. PMID 20724891
- [Background] Delannoy B, Wallet F, Maucort-Boulch D, Page M, Kaaki M, Schoeffler M, Alexander B, Desebbe O. Applicability of Pulse Pressure Variation during Unstable Hemodynamic Events in the Intensive Care Unit: A Five-Day Prospective Multicenter Study. Crit Care Res Pract. 2016;2016:7162190. doi: 10.1155/2016/7162190. Epub 2016 Mar 31. PMID 27127648